CLINICAL TRIAL: NCT06944301
Title: Comparison of Myocardial Injury After Noncardiac Surgery (MINS) Incidence in Supine vs. Prone Positioning During Percutaneous Nephrolithotomy (PNL)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, medical doctor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 3211789
Record Dates: First submitted 2025-04-15; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: MINS; Myocardial Injury After Noncardiac Surgery; Myocardial Injury After Noncardiac Surgery (MINS); Renal Calculi; Renal Stones; Percutaneous Nephrolithotomy (PNL); Nephrolithiasis
Keywords: MINS; PNL; percutaneous nephrolithotomy; Myocardial Injury after Noncardiac Surgery; prone; supine
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Deception | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine PNL (Other): Patients undergoing PNL in the supine position.
  Interventions: Diagnostic Test: blood sampling
- Prone PNL (Other): Patients undergoing PNL in the prone position.
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — measuring troponine preoperative and postoperative first and second day

SUMMARY:
This prospective cohort study aims to compare the incidence of Myocardial Injury after Noncardiac Surgery (MINS) in patients undergoing percutaneous nephrolithotomy (PNL) for kidney stones in supine versus prone positioning. MINS is defined as an elevated postoperative troponin level (≥0.03 ng/mL) within 48 hours after surgery. Approximately 400 patients will be enrolled, with 200 patients in each positioning group (supine and prone). The primary outcome is the incidence of MINS, assessed through troponin measurements and electrocardiogram (ECG) findings. Secondary outcomes include intraoperative complications, duration of surgery, and postoperative recovery metrics. The study seeks to determine whether surgical positioning impacts MINS risk, potentially guiding safer surgical practices.

DETAILED DESCRIPTION:
Myocardial Injury after Noncardiac Surgery (MINS) is a significant perioperative complication associated with increased morbidity and mortality. This study investigates whether surgical positioning (supine vs. prone) during percutaneous nephrolithotomy (PNL) influences the incidence of MINS. Patients aged 18 years and older undergoing PNL for kidney stones will be enrolled in a prospective cohort study at [Institution Name]. Exclusion criteria include pre-existing cardiovascular disease, elevated baseline troponin levels, or major intraoperative complications. Approximately 400 patients will be divided into two groups based on surgical positioning: 200 in the supine group and 200 in the prone group. Troponin levels will be measured preoperatively and at 24 and 48 hours postoperatively, with MINS defined as a troponin T level ≥0.03 ng/mL. Electrocardiograms (ECGs) will be performed to detect ischemic changes. Secondary outcomes include intraoperative hypotension, surgical duration, and postoperative hospital stay. Data will be analyzed using chi-square tests and logistic regression to adjust for confounders such as age, comorbidities, and surgical duration. The study aims to provide evidence on the impact of positioning on MINS, potentially informing safer surgical protocols for PNL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years.
* Patients undergoing percutaneous nephrolithotomy (PNL) for kidney stones.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Known coronary artery disease, heart failure, or other significant cardiovascular conditions.
* Elevated preoperative troponin levels (≥0.03 ng/mL).
* Major intraoperative complications (e.g., severe bleeding requiring transfusion).
* Inability to comply with study procedures.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Myocardial Injury after Noncardiac Surgery (MINS) | Up to 48 hours post-surgery
  Proportion of patients with postoperative troponin T levels ≥0.03 ng/mL within 48 hours after PNL, confirmed by ECG findings if ischemic changes are present.

SECONDARY OUTCOMES:
Surgical Duration | During surgery.
  Time from incision to closure (in minutes).
Postoperative Hospital Stay | From surgery to discharge.
  Duration of hospital stay after surgery (in days).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient privacy. Aggregated data may be published in scientific journals.

REFERENCES:
- [Background] Saha S, Dua A. Stochastic Lindemann kinetics for unimolecular gas-phase reactions. J Phys Chem A. 2013 Aug 22;117(33):7661-9. doi: 10.1021/jp402675s. Epub 2013 Aug 13. PMID 23879409
- [Background] Li L, Quang TS, Gracely EJ, Kim JH, Emrich JG, Yaeger TE, Jenrette JM, Cohen SC, Black P, Brady LW. A Phase II study of anti-epidermal growth factor receptor radioimmunotherapy in the treatment of glioblastoma multiforme. J Neurosurg. 2010 Aug;113(2):192-8. doi: 10.3171/2010.2.JNS091211. PMID 20345222
- [Background] Preston GC, Keene ON, Palmer JL. The effect of ondansetron on the pharmacokinetics and pharmacodynamics of temazepam. Anaesthesia. 1996 Sep;51(9):827-30. doi: 10.1111/j.1365-2044.1996.tb12610.x. PMID 8882243
- [Background] Edward GM, Das SF, Elkhuizen SG, Bakker PJ, Hontelez JA, Hollmann MW, Preckel B, Lemaire LC. Simulation to analyse planning difficulties at the preoperative assessment clinic. Br J Anaesth. 2008 Feb;100(2):195-202. doi: 10.1093/bja/aem366. PMID 18211993
- [Background] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- [Background] Chretien AE, Gagnon-Arsenault I, Dube AK, Barbeau X, Despres PC, Lamothe C, Dion-Cote AM, Lague P, Landry CR. Extended Linkers Improve the Detection of Protein-protein Interactions (PPIs) by Dihydrofolate Reductase Protein-fragment Complementation Assay (DHFR PCA) in Living Cells. Mol Cell Proteomics. 2018 Feb;17(2):373-383. doi: 10.1074/mcp.TIR117.000385. Epub 2017 Dec 4. PMID 29203496
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280